CLINICAL TRIAL: NCT04686448
Title: Propofol-Ketamine (Ketofol) Versus Propofol-Fentanyl (Fenofol) as Procedural Sedation for Unilateral Open Carpal Tunnel Release Under Local Anesthesia
Brief Title: Ketofol Versus Fenofol as Procedural Sedation for Carpal Tunnel Release
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mahmoud Abd Allah Zakzouk, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6556
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Procedural Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol-ketamine (Active Comparator): patients will receive IV ketofol (0.5 mg/kg ketamine and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4
  Interventions: Drug: propofol-ketamine
- propofol-fentanyl (Active Comparator): patients will receive IV fenofol (1 µg/kg fentanyl and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4
  Interventions: Drug: propofol-fentanyl

INTERVENTIONS:
Drug: propofol-ketamine — patients will receive IV ketofol (0.5 mg/kg ketamine and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4
  Other Names: ketofol
  Arms: propofol-ketamine
Drug: propofol-fentanyl — patients will receive IV fenofol (1 µg/kg fentanyl and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4
  Other Names: fenofol
  Arms: propofol-fentanyl

SUMMARY:
There are different methods of anesthesia for CTR surgery. Procedural sedation will allow rapid recovery and fewer complications than regional or general anesthesia (GA).

Attempts have been made in the past to use additives with propofol to reduce its dose. Ketofol (ketamine/propofol combination) was used for procedural sedation and analgesia. Ketamine and propofol administered in combination have offered effective sedation for spinal anesthesia and for gynecologic, ophthalmologic, and cardiovascular procedures in all age groups. The opposing hemodynamic and respiratory effects of each drug may enhance the utility of this drug combination, increasing both safety and efficacy and allowing reduction in the dose of propofol required to achieve sedation.

Propofol alone had a significantly greater number of apnea with desaturation (SpO2 < 90%) episodes. Further, it has been shown that during colonoscopies, propofol in combination with fentanyl provided similar patient satisfaction with shorter recovery times even at lower depths of sedation as compared to propofol. The addition of fentanyl to propofol has been shown to result in better operator feasibility with no difference in recovery time, cognitive impairment, or complications as compared to the use of propofol only for sedation.

DETAILED DESCRIPTION:
Sample size: assuming that the sedation using modified Ramasy sedation score was 6±0.01 in ketofol group versus 5.38±0.87 in fenofol group so the sample will be 56 patients, 28 patients in each group using OPENEPI at power 80 and CI 95 A computer-generated randomization table divided patients into 2 equal groups.

* Group (K) (n=28): patients will receive IV ketofol (0.5 mg/kg ketamine and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4.
* Group (F) (n=28): patients will receive IV fenofol (1 µg/kg fentanyl and 1 mg/kg propofol) as bolus injection over 5 minutes in the same syringe then infusion of 0.05 mg/kg/min propofol increased or decreased rate of infusion according to achieve sedation response by modified Ramasy sedation score of ≤ 4.

The depth of sedation will be assessed by modified Ramsay sedation

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-55 years old.
* Sex: both sex (males or females).
* Physical status: ASA I & II.
* BMI: 25-30 kg/m2.
* Type of operation: elective unilateral CTR under local anesthesia.
* Written informed consent from the patient.
* Cooperative patient.

Exclusion Criteria:

* Patient refusal.
* Altered mental status.
* Patients with known history of allergy to study drugs.
* Severe hepatic, renal, Cardiovascular and respiratory diseases.
* Patients on regular sedative or pain killer medications.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
depth of sedation | from drug injection up to 15 minutes till modified Ramsay sedation scale ≤ 4
  assessed by Modified Ramsay sedation scale. Score Modified Ramsay Sedation Scale Score
  1. Awake and alert, minimal or no cognitive impairment
  2. Awake but tranquil, purposeful responses to verbal commands at conversational level
  3. Appears asleep, purposeful responses to verbal commands at conversational level
  4. Appears asleep, purposeful responses to verbal commands but at louder than usual conversational level, requiring light glabellar tap, or both
  5. Asleep, sluggish purposeful responses only to loud verbal commands, strong glabellar tap, or both
  6. Asleep, sluggish purposeful responses only to painful Stimuli
  7. Asleep, reflex withdrawal to painful stimuli only (no purposeful responses)
  8. Unresponsive to external stimuli, including pain interpretation: score 1= minimal sedation score 2-4=moderate sedation score 5-7=deep sedation score 8=anesthesia

SECONDARY OUTCOMES:
recovery time | up to 30 minutes postoperative
  The time from discontinuation of infusion drug to first response to verbal command
• The total duration of post-anesthesia care unit (PACU) stay (The time from arrival to the PACU to discharge to the ward) according to modified Aldrete score 9 | up to 1 hour postoperative
  Modified Aldert score. Assessment items Condition Grade Activity, able to move, voluntarily or on command 4 extremities 2 2 extremities 1 No 0
  Breathing Able to breathe deeply & cough freely 2 Dyspnea, shallow or limited breathing 1 Apnea 0
  Consciousness Fully awake 2 Arousable on calling 1 Unresponsive 0 Circulation (BP) ±20% of pre-anesthesia level 2
  * 20% to 49% of pre-anesthesia level 1
  * 50% of pre-anesthesia level 0
  SPO2 Maintains SpO2 >92% in ambient air 2 Maintain SpO2 >90% with O2 1 Maintain SpO2 <90% with O2 0
  • Patient having a score of 9 or higher is discharged
Total propofol consumption by mg | from the start of drug injection till discontinuation of propfol infusion about 1 hour
  intraoperatice total propofol consumption by mg
number of participants with intraoperative complications such as hypotenstion, bradycardia and hypoxia | from the start of drug injection till end of surgery about 1 hour
  Intraoperative Complications such as hypotension (a decrease in mean arterial pressure 20% from base line mean arterial pressure, it will be treated with intravenous fluids and incremental doses of ephedrine), bradycardia (a decrease in heart rate 20% from base line heart rate, it will be treated with atropine) and hypoxia (a decrease in O2 saturation below 92%) will be treated with increasing O2 flow
number of participants with postoperative complications such as postoperative nausea and vomting | within 12 hours postoperative
  number of participants with postoperative complications such as postoperative nausea and vomting

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Zakzouk, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt